CLINICAL TRIAL: NCT06739499
Title: Bern, Get Ready (BEready) Population-based Cohort Study for Pandemic Preparedness: Main Study
Brief Title: Bern, Get Ready (BEready) Cohort Study for Pandemic Preparedness
Acronym: BEready
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Stiftung Vinetum (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-02290
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pandemic, COVID-19; Infections; Zoonoses; Epidemic Disease; Respiratory Tract Infections
Keywords: One Health; Pandemic preparedness; Community engagement
MeSH Terms: conditions — COVID-19; Infections; Zoonoses; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The BEready project aims to find out how people in the Canton of Bern can be helped to be more prepared for the next pandemic. BEready wants to understand how infections spread among people as well as between people and animals. BEready wants to find out how social and environmental factors can influence the transmission or catching of infectious diseases. BEready wants to better understand how households and their pets in the Canton of Bern were and continue to be affected by the coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
The overall aim is to establish BEready as a 'pandemic preparedness cohort', a cohort with a well-characterised study population of households, which has an infrastructure to conduct studies about infectious diseases, and which can be rapidly mobilised to respond to a new pandemic. BEready aims to understand the epidemiology and transmission of infectious diseases (particularly viral respiratory pathogens) in households including pets in the canton of Bern, and to engage diverse communities in efforts to strengthen pandemic preparedness.

The objectives are:

* to study the distribution and timing of infectious diseases and transmission patterns of circulating infectious diseases, both between individuals and at the human-animal interface (One Health)
* to study social (e.g. gender, affective polarisation) and environmental factors (e.g. climate change), which may affect transmission or acquisition of infectious diseases;
* to understand how households, including their pets, in the canton of Bern have been and will be affected by COVID-19; and
* to engage diverse communities in ongoing efforts to strengthen pandemic and public health literacy, and to prepare for the public health response to a new pandemic.

ELIGIBILITY:
Inclusion criteria for adults and children:

* Informed consent
* Residence (average of more than 3 days/week) in a private household in the canton of Bern where at least one member aged 18 agreed to take part.
* For adults, children aged 14 years or older, and parents/legal guardians: internet connection (Wi-Fi, fixed or on a mobile phone) and personal email address.
* For adults, children aged 11 years or older, and parents/legal guardians: able to understand, speak, read and write German, French and/or English.

Inclusion criteria for household pets: Pets of eligible household members with the consent of their owners.

Exclusion criteria for adults and children: Currently planned move outside the canton of Bern

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: BEready will include a spectrum of the Bernese population living in private households, including adults, children and pets. A private household is defined as a person living alone or group of persons living in the same dwelling.
  The study population for the BEready cohort will be enrolled from different sources in the source population of the canton of Bern. BEready aims to enrol around 1,500 households in total from:
  * Households already participating in the BEready pilot study
  * A random selection of households in Bern using the cantonal residents' register
  * Volunteer households from the general public
Sampling Method: Probability Sample
Enrollment: 2157 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2100-12-31 (Estimated); Study Completion 2100-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate among the randomly sampled participants | Baseline
  Percentage agreeing to take part, divided by the number invited, by age and sex (study level)
Attendance of follow up visits (to derive factors associated with research participation) | At every annual follow-up for up to 100 years
  Percentage of completed questionnaire (study level)
Incidence of respiratory virus detection in symptomatic persons | At the end of a 12 months period
  Test positivity: percentage of nasal swab samples with a positive result for specific respiratory viruses among all viruses detected amongst those reporting disease events cumulatively by the end of one year; incidence rate for any detected virus and for specific viruses: number of nasal swab samples with a positive result per 100 person years of follow-up (individual level, infection-related)
Seroprevalence of antibodies to respiratory viruses | At baseline and annually thereafter for up to 100 years
  Proportion of serum samples with antibodies to specific respiratory viruses (individual level, infection-related)
Incidence of co-infection/co-colonisation at the pet/owner interface | Throughout follow-up for up to 100 years
  Proportion of serum samples with antibodies to specific parasites (individual level, infection-related)
Incidence of animal diseases diagnosed through syndromic surveillance | Throughout follow-up for up to 100 years
  Based on each case definition, e.g. febrile illness, incidence of syndromic diagnoses by month (individual level, infection-related)
Prevalence of post-acute viral symptoms | At baseline and annually thereafter for up to 100 years
  Individual level, infection-related
Gender roles | At all timepoints for up to 100 years
  Gender is a cross-cutting theme. Associations with gender measured by questionnaire will be examined for all endpoints (individual level, personal, social, demographic).
Number of daily social contacts | At baseline and annually thereafter for up to 100 years
  Numbers of social contacts between humans, according to age group and location (individual level, personal, social, demographic)
Affective polarisation | At baseline
  Mean and standard deviation of Likert scale scores (individual level, personal, social, demographic)
Knowledge of pandemic preparedness | At baseline
  Knowledge measured by questionnaire. Summary of the survey data (individual level, personal, social, demographic)
Knowledge of vector-borne diseases | At baseline
  Knowledge measured by questionnaire. Summary of the survey data (individual level, personal, social, demographic)
Experienced marginalisation | At baseline
  Experience measured by questionnaire. Summary of the survey data (individual level, personal, social, demographic)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Low, Prof. Dr. med., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Upon request

REFERENCES:
- See also: BEready Cohort study website — https://www.beready.unibe.ch/index_eng.html